CLINICAL TRIAL: NCT06055738
Title: An Exploratory Clinical Study of Zimberelimab Combined With Albumin-bound Paclitaxel and Cisplatin in Neoadjuvant Treatment of Locally Advanced Cervical Cancer
Brief Title: Zimberelimab Combined With Albumin-bound Paclitaxel and Cisplatin in Neoadjuvant Treatment of LACC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TangduH-1
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Locally Advanced Cervical Cancer
MeSH Terms: interventions — zimberelimab; Albumin-Bound Paclitaxel; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zimberelimab combined with albumin-bound paclitaxel and cisplatin (Experimental): Zimberelimab combined with albumin-bound paclitaxel and cisplatin in neoadjuvant treatment of locally advanced cervical cancer
  Interventions: Drug: Zimberelimab; Drug: Albumin-bound Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Zimberelimab — 240mg,d1,iv,Q21D
  Other Names: GLS-010
Drug: Albumin-bound Paclitaxel — 260mg/m2,d1,iv,Q21D
  Other Names: Paclitaxel
Drug: Cisplatin — 75mg/m2,d1,iv,Q21D
  Other Names: CDDP

SUMMARY:
This is a prospective, single arm, phase II clinical study to evaluate the efficacy and safety of Zimberelimab combined with albumin-bound paclitaxel and cisplatin as neoadjuvant therapy for locally advanced cervical cancer.

DETAILED DESCRIPTION:
This study will enroll patients with IB3 and IIA2 locally advanced cervical cancer who received three cycles of neoadjuvant Zimberelimab combined with albumin-bound paclitaxel and cisplatin to evaluate the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in clinical research.
2. Age ≥18 years old, female.
3. Squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the cervix confirmed by histology/cytology.
4. Previously untreated locally advancedcervical cancer (2018 FIGO stage IB3, IIA2) .
5. At least one measurable lesion was suitable for target lesion according to RECIST v1.1 .
6. Within 14 days before the first treatment, the major organ functions were basically normal.
7. Eastern Cooperative Oncology Group (ECOG) performance status score 0-1;
8. Subjects agree to provide sufficient tumor tissue samples for PD-L1 expression detection;
9. If hepatitis B surface antigen (HBsAg) is positive and/or hepatitis B core antibody (HBcAb) is positive, hepatitis B virus DNA (HBV DNA) is detected, HBV DNA < 104 copies /ml or < 2000IU/mL can be enrolled. Or those who had received antiviral therapy for at least 4 weeks before the first dose of study drug and were willing to continue antiviral therapy during the study were eligible for enrollment. Those with HCV antibody positive should be excluded.
10. Subjects of childbearing age and their sexual partners agreed to consent to contraceptive use after signing an informed consent form, during treatment and for at least 6 months after the last dose of the study intervention.

Exclusion Criteria:

1. Patients with active autoimmune disease or a history of autoimmune disease.
2. Previous history of allogeneic hematopoietic stem cell transplantation or organ transplantation (except corneal transplantation).
3. Use of immunosuppressive drugs within 14 days prior to treatment, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroids (i.e., not more than 10 mg/ day of prednisolone or another corticosteroid at the physiological dose of the drug).
4. Previous treatment with anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, anti-CD137 antibody, or anti-lymphocyte antigen 4 (CTLA-4) antibody.
5. Arterial or venous thromboembolic events within the previous 6 months, including myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic attack, pulmonary embolism, deep vein embolism or any other major thromboembolism, implantable venous access port or catheter-derived thrombosis, or superficial venous thrombosis. Except for patients with stable thrombus after conventional anticoagulant therapy, prophylactic use of low-dose low molecular weight heparin was allowed.
6. Previous history of gastrointestinal perforation, gastrointestinal fistula, genital fistula (such as vesicovaginal fistula, urethrovaginal fistula, vesicovaginal fistula, etc.); Patients were allowed if the perforation or fistula had been treated with diversion surgery, resection, or repair, and the disease was recovered or relieved as judged by the investigator.
7. Symptomatic congestive heart failure (New York Heart Association class II-IV) Arrhythmias with poorly controlled symptoms.
8. Active pulmonary tuberculosis, receiving anti-tuberculosis treatment.
9. Interstitial lung disease.
10. Severe infections that are active or poorly controlled clinically. Severe infection within 3 weeks before treatment, including but not limited to patients hospitalized for complications of infection, bacteremia, or severe pneumonia.
11. Central nervous system metastasis, leptomeningeal metastasis, spinal cord compression, or leptomeningeal disease.
12. Human immunodeficiency virus (HIV) infection, known syphilis infection.
13. Have received live vaccine within 4 weeks of the first use of the experimental drug, or plan to receive live vaccine during the study.
14. Known or suspected allergy to the trial drug or any drug related to the trial.
15. Pregnant or lactating women.
16. There were other conditions deemed by the investigator to be inappropriate for enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-09 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3-4 months
  Objective response rate based on RECIST v1.1, ORR was defined as the ratio of best complete response (CR) and partial response (PR) recorded from the start of treatment to the preoperative evaluation

SECONDARY OUTCOMES:
Complete pathological response (pCR) | one year
  Complete pathological response (pCR) was defined as the proportion of all surgical patients in whom no viable tumor cells were found in the resected specimen.
Major Pathological Response (MPR) | one year
  Major pathological response (MPR) was defined as the proportion of patients with ≤10% residual viable tumor cells in the resected specimen among all surgical patients.
R0 resection rate | one year
  R0 resection rate: defined as the proportion of patients undergoing surgical excision who had a negative margin of surgical specimens
Event-free survival (EFS) | three years
  Event-free survival (EFS) was defined as the time from the start of treatment to the first occurrence of any of the following events: disease progression beyond surgical treatment, local or distant recurrence, death from any cause, etc.
Overall survival (OS) | three years
  Overall survival (OS) : defined as the time between the initiation of treatment and death from any cause.
Adverse Events | three years
  Based on NCI-CTC AE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Hongxi Zhao, PhD, Principal Investigator — Tangdu Hospital-Air Force Medical University
Locations (1):
- Hongxi Zhao, Xi'an, Shaanxi, China